CLINICAL TRIAL: NCT06258928
Title: Early Mobilisation of the Distal Radius Fracture Isokinetic and Functional Evaluation
Brief Title: Early Mobilisation of the Distal Radius Fracture
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Magdalena Kolasińska, Principal Investigator, Józef Piłsudski University of Physical Education
Other Study IDs: Radius Fracture
Record Dates: First submitted 2024-02-03; First posted 2024-02-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Secondary Prevention
Keywords: distal radius fracture; early therapy; exercise therapy
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a distal radius fracture: Functional examination included evaluating range of motion (ROM), grip strength, and isokinetic evaluation of force moments (Biodex) for wrist flexion, extension, forearm pronation, and forearm supination. Michigan's questionnaire and the Disability of the Arm, Shoulder, and Hand (DASH) questionnaire were used to subjectively evaluate the effects of therapy.
  Interventions: Diagnostic Test: Functional examination

INTERVENTIONS:
Diagnostic Test: Functional examination — Compared to nonoperated limb, after 6 months of early rehabilitation.

SUMMARY:
The goal of this clinical trial is to demonstrate the effectiveness of early therapy in 14 patients with a distal radius fracture DRF resulting from injury, as the study group. Assess hand function of patients who underwent surgical repair of distal radius fractures using the open reduction internal fixation method (ORIF), compared to their nonoperated limb, after 6 months of early rehabilitation.

The main questions it aims to answer are:

1. Significantly faster recovery of independence from daily activities by the patient.
2. For economic reasons, patients often expect to return to work as soon as possible.

Participants will be subjected to functional examination to assess hand function of patients who underwent surgical repair of distal radius fractures using the open reduction internal fixation method.

ELIGIBILITY:
Inclusion Criteria:

* age range 18-60 years
* distal radius fracture
* ORIF procedure
* hand stabilisation plate (Medartis)

Exclusion Criteria:

* delayed rehabilitation protocol
* algodystrophy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with a distal radius fracture DRF resulting from injury
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
DASH -Disability of the Arm, Shoulder, and Hand | 1 day
  questionnaire assesses upper limb disability and consists of 30 questions in the general section and an additional work module with 4 questions and a sport/instrument playing module with 4 questions. Assess symptoms and the inability to perform certain activities based on health status.
ROM - range of motion | 1 day
  Flexion, extension of the wrist, supination and pronation of the forearm using a 15 cm stainless steel Saehan finger goniometer
Grip strength | 1 day
  Using a hydraulic handgrip dynamometer by Saehan according to the procedure to measure grip strength
Isokinetic evaluation | 1 day
  Isokinetic evaluation of force moments of the biceps and triceps, and the muscles responsible for supination and pronation of the forearm using the Biodex System 4 Pro (Biodex, USA) dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Terapia Ręki Magda Kolasińska, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No